CLINICAL TRIAL: NCT00664859
Title: A 12-Month, Open-Label, Extension Study of the Safety and Efficacy of LCP-AtorFen in Subjects With Dyslipidemia
Brief Title: 12-Month, Open-Label, Extension Study of LCP-AtorFen in Dyslipidemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCP-AtorFen-2001-1X
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Dyslipidemia
Keywords: LCP-AtorFen; Non-HDL cholesterol; Triglycerides; HDL cholesterol; LDL cholesterol; Atorvastatin; Fenofibrate
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): Open-label LCP-AtorFen
  Interventions: Drug: LCP-AtorFen

INTERVENTIONS:
Drug: LCP-AtorFen — All subjects will be assigned to receive open-label LCP-AtorFen combination therapy for 52 weeks. Subjects will take a single oral dose of study drug in the evening without regard to meals.
  Other Names: atorvastatin and fenofibrate combination therapy

SUMMARY:
The current study is designed to test the long-term (12-month) safety and efficacy of LCP-AtorFen, a combination of atorvastatin and fenofibrate, in patients with dyslipidemia

DETAILED DESCRIPTION:
POPULATION:

Subjects with mixed dyslipidemia (non-HDL cholesterol > 130 mg/dL and TG ≥ 150 mg/dL and ≤ 500 mg/dL) who completed the double-blind study (LCP-AtorFen-2001; NCT00504829), met the enrollment criteria (all of the inclusion criteria and none of the exclusion criteria), and elected to enter the open-label extension study.

STUDY DESIGN AND DURATION:

This is a 52-week, open-label, single-treatment arm with 8 visits (Weeks 0, 4, 8, 12, 24, 36, 48 and 52). A maximum of approximately 200 subjects will enter this open-label safety and efficacy extension study from the LCP AtorFen-2001 double-blind study. All subjects enrolled in this study will receive open-label LCP-AtorFen combination therapy. Visit 1 of the extension study corresponds to the last visit of the double-blind study (Visit 6 or Week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has successfully completed the double-blind study (LCP-AtorFen-2001; NCT00504829).
2. Subject has confirmed his or her willingness to participate in this study after being informed of all aspects of the study by voluntarily signing and dating an informed consent form in accordance with Good Clinical Practice (GCP).

Exclusion Criteria:

1. Study drug compliance <70% in the double-blind study.
2. Any ongoing serious adverse event, or any ongoing non-serious moderate or severe adverse event from the double-blind study that is rated as possibly, probably or definitely related to study drug.
3. Resting blood pressure >/=160 mm Hg systolic and/or >/=100 mm Hg diastolic.
4. Symptoms of unexplained muscle pain, tenderness or weakness (i.e., signs indicative of possible myopathy), or any diagnosis of myopathy or rhabdomyolysis.
5. Any clinically significant change in physical exam or electrocardiogram from Visit 2 to Visit 6 of the double-blind study.
6. Any clinically significant change from Visit 1 to Visit 6 of the double-blind study in medical history including, but not limited to: a diagnosis of insulin-dependent diabetes mellitus (DM); poorly controlled DM; poorly controlled hypertension; significant renal, pulmonary, hepatic, biliary, or gastrointestinal disease; cancer (except non-melanoma skin cancer); and epilepsy.
7. Unwilling to abstain from medications, supplements, ingredients and herbal therapies that were excluded in the double-blind study and continue to be excluded in the open-label study.
8. Women who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential (not surgically sterilized between menarche and menopause) who are not using a medically approved method of contraception.
9. Other exclusion conditions might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Geohas, MD, Principal Investigator — Radiant Research; Dennis McCluskey, MD, Study Director — Radiant Resaerch; Harry Geisberg, MD, Study Director — Radiant Research; Chivers Woodruff, Jr, MD, Study Director — Radiant Research; Michael Noss, MD, Study Director — Radiant Research; Michele Reynolds, MD, Study Director — Radiant Research; James Zavoral, MD, Study Director — Radiant Research; Randall Severance, MD, Study Director — Radiant Research; Stephen Halpern, MD, Study Director — Radiant Research; Linda Murray, MD, Study Director — Radiant Research; Eduardo Cuevas, MD, Study Director — Radiant Research; Cynthia Strout, MD, Study Director — Coastal Carolina Research; Mark Kipnes, MD, Study Director — Diabetes and Glandular Research Center, Inc.
Locations (1):
- Radiant Research, 515 N State St, Suite 2700, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 192 subjects who completed the double-blind (DB) period, 140 rolled over into the extension study and received at least one dose of open-label (OL) study drug to form the safety population.
Groups:
- LCP-AtorFen 40/100 mg: Subjects randomized to LCP-AtorFen 40/100 mg/day in the DB portion of the study
- Atorvastatin 40 mg: Subjects randomized to Atorvastatin 40 mg/day in the DB portion of the study
- Fenofibrate 145 mg: Subjects randomized to Fenofibrate 145 mg/day in the DB portion of the study
Period: Overall Study
Arm/Group | LCP-AtorFen 40/100 mg | Atorvastatin 40 mg | Fenofibrate 145 mg
Started | 51 | 45 | 44
Completed | 34 | 35 | 23
Not Completed | 17 | 10 | 21
Not completed — Adverse Event | 2 | 1 | 3
Not completed — DB Study (LCP-AtorFen-2001) AE | 6 | 4 | 4
Not completed — Noncompliance with protocol | 1 | 0 | 4
Not completed — Laboratory abnormality | 2 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 1 | 3
Not completed — Lost to Follow-up | 2 | 2 | 1
Not completed — Other | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- LCP-AtorFen 40/100mg; Atorvastatin 40 mg; Fenofibrate 145 mg: Data presented by previous double-blind study assignment
- Total: Total of all reporting groups
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40 mg | Fenofibrate 145 mg | Total
Number analyzed (Participants) | 51 | 45 | 44 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.86) | 55.6 (9.03) | 57.2 (11.23) | 55.7 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 17 | 55
  Male | 33 | 25 | 27 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Amer. Indian /Alaskan | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Black/African | 3 | 3 | 1 | 7
  Hawaiian/Other | 0 | 0 | 0 | 0
  White | 46 | 38 | 42 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change in Non-HDL Cholesterol, HDL Cholesterol, TG Levels From Baseline to End of Treatment
Description: Mean percent changes in non-HDL cholesterol, HDL cholesterol, TG levels from the double-blind (DB) baseline (Week 0) to end-of-treatment (Week 52), and from the open-label (OL) baseline (week 12 of DB study) to end of treatment (Week 52)
Time Frame: 52 weeks from DB baseline and 40 weeks from OL baseline
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40 mg | Fenofibrate 145 mg
Number analyzed (Participants) | 51 | 44 | 43
percent change
  Non-HDL cholesterol, change from DB baseline | -48.2 (13.58) | -43.6 (18.18) | -42.0 (20.49)
  Non-HDL cholesterol change from OL baseline | 2.6 (22.39) | 2.8 (33.67) | -29.6 (26.92)
  Triglycerides change from DB baseline | -53.1 (25.31) | -51.2 (23.23) | -42.1 (29.96)
  Triglycerides change from OL baseline | 11.4 (65.36) | -19.1 (40.42) | -5.2 (53.27)
  HDL cholesterol change from DB baseline | 22.1 (21.7) | 16.3 (18.67) | 17.5 (20.21)
  HDL cholesterol change from OL baseline | 2.1 (16.9) | 10.1 (17.77) | -2.4 (15.4)

2. Secondary Outcome: Change in LDL Cholesterol, VLDL, Total Cholesterol, Apo A-1, and Apo B From Baseline to End of Treatment
Description: Mean percent changes in LDL cholesterol, VLDL, total cholesterol, Apo A-1, and Apo B from the double-blind (DB) baseline (Week 0) to end-of-treatment (Week 52), and from the open-label (OL) baseline (week 12) to end-of-treatment (Week 52)
Time Frame: 52 weeks from DB baseline and 40 weeks from OL baseline
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40 mg | Fenofibrate 145 mg
Number analyzed (Participants) | 51 | 44 | 43
Percent change
  LDL-C change from DB baseline | -44.8 (15.92) | -39.3 (20.04) | -40.9 (22.0)
  LDL-C change from OL baseline | 2.1 (25.09) | 14 (36.29) | -33.6 (24.26)
  VLDL-C change from DB baseline | -53.6 (23.98) | -51.1 (23.07) | -42.0 (29.94)
  VLDL-C change from OL baseline | 12.7 (69.42) | -18.7 (39.97) | -5.5 (51.98)
  Total-C change from DB baseline | -36.5 (11.07) | -33.8 (14.6) | -32.8 (16.08)
  Total-C change from OL baseline | 1.5 (12.95) | 4.6 (24.54) | -24.4 (19.04)
  Apo A-1 change from DB baseline | 3.2 (13.21) | 1.0 (9.88) | 0.4 (12.5)
  Apo-A-1 change from OL baseline | -1.4 (8.11) | 1.9 (13.62) | -5.1 (11.36)
  Apo B change from DB baseline | -42.4 (11.85) | -38.9 (16.26) | -36.8 (18.81)
  Apo B change from OL baseline | 3.1 (17.69) | -1.5 (25.14) | -25.5 (21.59)

ADVERSE EVENTS:
Arm/Group | LCP-AtorFen 40/100mg | Atorvastatin 40 mg | Fenofibrate 145 mg
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/45 | 3/44
Other Adverse Events (participants affected / at risk) | 12/51 | 21/45 | 21/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCP-AtorFen 40/100mg (N=51) | Atorvastatin 40 mg (N=45) | Fenofibrate 145 mg (N=44)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fracture treatment (Injury, poisoning and procedural complications) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 0 | 1
Elevated ALT (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCP-AtorFen 40/100mg (N=51) | Atorvastatin 40 mg (N=45) | Fenofibrate 145 mg (N=44)
Diarrhoea (Gastrointestinal disorders) | 1 | 6 | 1
Nasopharyngitis (Infections and infestations) | 6 | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 4
Blood glucose increased (Endocrine disorders) | 1 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 3
Haematuria (Renal and urinary disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study is a multicenter collaborative investigation and the clinical trial results are to be published as a collaborative manuscript. Authorship will reflect varying levels of individual contribution to the study by the individual PI's.